## TITLE PAGE- STUDY PROTOCOL

| Manuscript Title: |
|---|
| Evaluation of Factors Influencing Antibiotic Use in RSV-Positive Infants: A Retrospective |
| Observational Study |
| Running Title: |
| RSV Antibiotic Use: Drivers and Cost |
| Authors: |
| Burcu Büşra Acar¹, Elif Böncüoğlu³, Şahika Şahinkaya², Elif Kıymet⁴,İlker Devrim², |
| Author Affiliations: |
| 1. Department of Pediatric Cardiology, Ege University Faculty of Medicine, Izmir, Türkiye |
| 2. Department of Pediatric Infectious Diseases, Dr. Behçet Uz Children's Hospital, Izmir, |
| Türkiye |
| 3. Department of Pediatric Infectious Diseases, Faculty of Medicine, Izmir Bakırçay University |
| Izmir, Türkiye |
| 4. Department of Pediatric Infectious Diseases, Faculty of Medicine, Izmir Demokrasi |
| University, Izmir, Türkiye |

| Corresponding Author: |
|---|
| Burcu Büşra Acar, MD |
| Ege University Faculty of Medicine, Department of Pediatric Cardiology, 35100 Bornova, Izmir, |
| Türkiye |
| Phone: +90 507 479 78 35 |
| E-mail: drburcubusraacar@gmail.com |
| Funding: |
| This study was not supported by any public or private institution. |
| Conflict of Interest: |
| The authors declare no conflict of interest. The datasets generated and/or analyzed during the |
| current study are available from the corresponding author on reasonable request. |
| Acknowledgements: |
| None. |
| Presentation at Meetings: |
| This study was presented as an oral presentation at the 2nd International Behçet Uz Pediatric |
| Congress held in İzmir, Turkey, on September 22–24, 2022. |
| NCT Number: Pending |

Document Date: May 10, 2025